CLINICAL TRIAL: NCT03501836
Title: Performance Evaluation Study of a Six Electrode (8 Lead) Wireless Handheld ECG Recording Device With Four Lead Chest Extension Versus Conventional 12-lead ECG in Heart Patients
Brief Title: Wireless Handheld 8-lead ECG Device Performance in Heart Patients (Rapid Rhythm)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: Rapid Rhythm Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 160483; R04118 (Other: Central Manchester University Hospitals NHS Foundation Trust)
Record Dates: First submitted 2018-04-09; First posted 2018-04-18 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Atrial Fibrillation; Heart Murmurs
MeSH Terms: conditions — Atrial Fibrillation; Heart Murmurs

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rapid Rhythm Handheld 8-lead ECG Device (Experimental): Participants will have measurements taken with the 8 lead ECG system, which will be compared to the conventional standard care 12 lead ECG.
  Interventions: Device: Rapid Rhythm Handheld 8-lead ECG Device

INTERVENTIONS:
Device: Rapid Rhythm Handheld 8-lead ECG Device — We want to explore whether using 6 electrodes on the chest (as in the Rapid Rhythm Handheld 8-lead ECG device) can give the same diagnostic result to the standard 10 electrode (12-lead) ECG, which uses 6 chest electrodes plus 4 electrodes on the arms and legs.
  To do this we need to compare measurements taken with the 6 electrode (8 lead) study device to those taken with the gold-standard 10 electrode (12 lead) method.
  We want to find out whether the new equipment can detect the same heart rhythms as the standard method, so that ECG measurements might be made more quickly and easily in the future.

SUMMARY:
This study is designed to compare the performance of both 6 and 10 electrode ECGs from the handheld device with the conventional 12 lead ECG. As well as comparing the detection of atrial fibrillation, the study will also compare the detection of other heart problems and of normal heart rhythm.

DETAILED DESCRIPTION:
An Electrocardiogram (ECG) 6 electrode, wireless handheld device held on the chest is being developed to allow diagnosis of heart rhythm problems without the need for connecting electrodes to the chest, arms and legs as in a standard 10 electrode (referred to as a 12-lead) ECG measurement. A faster and simpler yet accurate method for acquiring ECG data may be useful in many healthcare settings, including screening for irregular heart rhythms such as Atrial Fibrillation (AF), which is a risk factor for stroke. The wireless 6 electrode device has an extension arm for the handset with 4 additional electrodes (also positioned on the chest) to give a full 12 lead ECG signal. This study is designed to compare the performance of both 6 and 10 electrode ECGs from the handheld device (used on the chest with the subject seated) with the conventional 12 lead ECG (used with electrodes on the chest, arms and legs with the subject lying down). As well as comparing the detection of atrial fibrillation, the study will also compare the detection of other heart problems and of normal heart rhythm. Adult patients attending the clinics at Central Manchester University Hospitals NHS Foundation Trust for an ECG assessment are eligible to participate in the study. A maximum of 500 patients will be recruited to the study in order to find the number of cases with Atrial Fibrillation required to properly compare the methods. A subset of patients with normal ECGs will have additional measurements with both methods whilst lying down, reclining at an angle and sitting upright to investigate any effects of body posture on chest based ECGs.

ELIGIBILITY:
Inclusion Criteria:

1. Patient attending an adult cardiology or anti-coagulation clinic appointment, at clinics at Central Manchester University Hospitals NHS Foundation Trust (including the Manchester Heart Centre).
2. Patients on cardiac wards 3 and 4.
3. Aged 18 years or above.
4. Male or Female.

Exclusion Criteria:

1. Aged less than 18 years.
2. Unable to give informed consent.
3. Does not wish to participate in the study.
4. Any patients with visible breaks to the skin, rashes or inflammation in the chest area on the day of the test
5. Bedridden or otherwise unable to transfer between chair and bed for both seated and supine measurements

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 271 (Actual)
Dates: Start 2017-01-24 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Capabilities of an 8 lead ECG system (Rapid Rhythm) - normal ECGs | 18 months
  The percentage of ECGs where a normal control ECG is matched by a normal RR ECG.
Capabilities of an 8 lead ECG system (Rapid Rhythm) - abnormal ECGs | 18 months
  The percentage of ECGs where abnormalities of the control ECG are matched by similar abnormalities of the RR ECG.

CONTACTS AND LOCATIONS:
Locations (1):
- Manchester University NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No